CLINICAL TRIAL: NCT00758836
Title: A Phase IIa Randomized, Double-Blind, Parallel-Group, Placebo and Active-Controlled, Clinical Trial to Study the Efficacy and Safety of MK0974 Co-administered With Ibuprofen or Acetaminophen in Patients With Migraine With or Without Aura
Brief Title: A Study to Test the Safety and Effectiveness of MK-0974 (Telcagepant) Co-administered With Ibuprofen or Acetaminophen in Patients With Migraines With or Without Aura (MK-0974-046)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0974-046; 2008_551 (Other: Merck Registration Number); CTRI/2009/091/000291 (Registry Identifier: CTRI)
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Ibuprofen; Acetaminophen; telcagepant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants take two placebo tablets and two placebo capsules, orally, at onset of migraine
  Interventions: Drug: placebo
- Telcagepant 280 mg +Ibuprofen 400 mg (Experimental): Participants take one telcagepant 280 mg tablet, one ibuprofen 400 mg tablet, and two placebo capsules, orally, at onset of migraine
  Interventions: Drug: ibuprofen; Drug: telcagepant
- Telcagepant 280 mg +APAP 1000 mg (Experimental): Participants take one telcagepant 280 mg tablet, one placebo tablet, and two 500-mg APAP capsules, orally, at onset of migraine
  Interventions: Drug: acetominophen; Drug: telcagepant
- Telcagepant 280 mg (Placebo Comparator): Participants take one telcagepant 280 mg tablet, one placebo tablet, and two placebo capsules, orally, at onset of migraine
  Interventions: Drug: telcagepant

INTERVENTIONS:
Drug: placebo
  Arms: Placebo
Drug: ibuprofen
  Arms: Telcagepant 280 mg +Ibuprofen 400 mg
Drug: acetominophen
  Other Names: N-acetyl-p-aminophenol (APAP)
  Arms: Telcagepant 280 mg +APAP 1000 mg
Drug: telcagepant
  Other Names: MK-0974
  Arms: Telcagepant 280 mg; Telcagepant 280 mg +APAP 1000 mg; Telcagepant 280 mg +Ibuprofen 400 mg

SUMMARY:
This study will test the safety and how effective telcagepant is when taken with ibuprofen or acetaminophen in participants with migraine with or without aura. The primary study hypothesis is that at least one drug combination is superior to telecagepant alone in the treatment of acute migraines.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* History of migraine with or without aura for more than 1 year with 1-8 moderate or severe migraine attacks per month in the 2 months prior to starting in the study
* Willing to stay awake for at least 2 hours after taking study drug
* Able to read, understand and complete questionnaires and diaries

Exclusion Criteria:

* Breast-feeding, pregnant, or plan to become pregnant during the study
* Not able to tell migraine attack from other headaches
* Older than 50 years of age at migraine onset
* Have more than 15 headache days per month or have taken medication for acute headache on more than 10 days per month in any of the 3 months before starting in the study
* History of gastric or small intestinal surgery
* History of heart attack, stroke, unstable angina, coronary artery bypass surgery or transient ischemic attack in the 3 months before starting in the study
* Currently participating or have participated in a study with in investigational compound or device in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2008-12-03 (Actual); Primary Completion 2009-08-24 (Actual); Study Completion 2009-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Hewitt DJ, Martin V, Lipton RB, Brandes J, Ceesay P, Gottwald R, Schaefer E, Lines C, Ho TW. Randomized controlled study of telcagepant plus ibuprofen or acetaminophen in migraine. Headache. 2011 Apr;51(4):533-43. doi: 10.1111/j.1526-4610.2011.01860.x. PMID 21457238
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0974-046&kw=0974-046&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Telcagepant 280 mg +Ibuprofen 400 mg | Telcagepant 280 mg +APAP 1000 mg | Telcagepant 280 mg
Started | 171 | 171 | 171 | 170
Treated | 147 | 145 | 133 | 138
Completed | 147 | 145 | 133 | 138
Not Completed | 24 | 26 | 38 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Telcagepant 280 mg +Ibuprofen 400 mg | Telcagepant 280 mg +APAP 1000 mg | Telcagepant 280 mg | Total
Number analyzed (Participants) | 171 | 171 | 171 | 170 | 683
Age, Customized [Number; unit: participants]
  <20 years | 4 | 0 | 3 | 3 | 10
  20-29 years | 34 | 43 | 32 | 33 | 142
  30-39 years | 33 | 47 | 37 | 53 | 170
  40-49 years | 58 | 51 | 49 | 51 | 209
  50-59 years | 32 | 19 | 42 | 23 | 116
  60-64 years | 4 | 6 | 6 | 2 | 18
  >=65 years | 6 | 5 | 2 | 5 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 139 | 149 | 145 | 583
  Male | 21 | 32 | 22 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pain Freedom at Two Hours Post-dose
Description: Pain severity was rated by the participants in a paper diary by grade; Grade 0 (no pain), Grade 1 (mild pain), Grade 2 (moderate pain), and Grade 3 (severe pain). Pain freedom was defined as a reduction in pain severity from moderate to severe migraine headache (Grade 2 or 3) to no pain (Grade 0).
Time Frame: 2 hours post-dose
Population: The Full Analysis Set (FAS) comprised participants who were treated and had a baseline assessment and at least one post-dose assessment up to or including the 2-hour time point. Missing data were imputed by using a Last Observation Carried Forward (LOCF) approach; baseline values were not carried forward to impute the missing post-treatment data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Telcagepant 280 mg +Ibuprofen 400 mg | Telcagepant 280 mg +APAP 1000 mg | Telcagepant 280 mg
Number analyzed (Participants) | 147 | 145 | 133 | 138
Percentage of Participants | 10.9 | 35.2 | 38.3 | 31.2
Statistical Analysis 1: Comparison: Placebo vs Telcagepant 280 mg +Ibuprofen 400 mg; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for independent binomial distribution stratified by baseline severity; Proportion difference = 24.5, 90% CI 2-sided [16.7 to 32.2]
Statistical Analysis 2: Comparison: Placebo vs Telcagepant 280 mg +APAP 1000 mg; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for independent binomal distribution stratified by baseline severity; Proportion difference = 27.7, 90% CI 2-sided [19.6 to 35.8]
Statistical Analysis 3: Comparison: Placebo vs Telcagepant 280 mg; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for independent binomal distribution stratified by baseline severity; Proportion difference = 20.4, 90% CI 2-sided [12.6 to 28.2]
Statistical Analysis 4: Comparison: Telcagepant 280 mg +Ibuprofen 400 mg vs Telcagepant 280 mg; Test type: Superiority or Other; p = 0.449, Miettinen and Nurminen; Miettinen and Nurminen method for independent binomal distribution stratified by baseline severity; Proportion differenece = 4.2, 90% CI 2-sided [-5.0 to 13.3]
Statistical Analysis 5: Comparison: Telcagepant 280 mg +APAP 1000 mg vs Telcagepant 280 mg; Test type: Superiority or Other; p = 0.182, Miettinen and Nurminen; Miettinen and Nurminen method for independent binomal distribution stratified by baseline severity; Proportion difference = 7.7, 90% CI 2-sided [-1.8 to 17.1]

2. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours Post-dose.
Description: Pain severity was rated by the participants in a paper diary by grade; Grade 0 (no pain), Grade 1 (mild pain), Grade 2 (moderate pain), and Grade 3 (severe pain). Pain relief was defined as a reduction in pain severity from moderate to severe migraine headache (Grade 2 or 3) to mild or none (Grade 1 or 0).
Time Frame: 2 hours post-dose
Population: The FAS comprised participants who were treated and had a baseline assessment and at least one post-dose assessment up to or including the 2-hour time point. Missing data were imputed by using a Last Observation Carried Forward (LOCF) approach; baseline values were not carried forward to impute the missing post-treatment data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Telcagepant 280 mg +Ibuprofen 400 mg | Telcagepant 280 mg +APAP 1000 mg | Telcagepant 280 mg
Number analyzed (Participants) | 147 | 145 | 133 | 138
Percentage of Participants | 30.6 | 71.0 | 69.9 | 65.2
Statistical Analysis 1: Comparison: Placebo vs Telcagepant 280 mg +Ibuprofen 400 mg; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for independent binomal distribution stratified by baseline severity; Proportion difference = 40.8, 90% CI 2-sided [31.9 to 49.0]
Statistical Analysis 2: Comparison: Placebo vs Telcagepant 280 mg +APAP 1000 mg; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for independent binomal distribution stratified by baseline severity; Proportion difference = 39.9, 90% CI 2-sided [30.5 to 48.5]
Statistical Analysis 3: Comparison: Telcagepant 280 mg +Ibuprofen 400 mg vs Telcagepant 280 mg; Test type: Superiority or Other; p = 0.265, Miettinen and Nurminen; Miettinen and Nurminen method for independent binomal distribution stratified by baseline severity; Proportion difference = 6.1, 90% CI 2-sided [-2.9 to 14.9]
Statistical Analysis 4: Comparison: Telcagepant 280 mg +APAP 1000 mg vs Telcagepant 280 mg; Test type: Superiority or Other; p = 0.362, Miettinen and Nurminen; Miettinen and Nurminen method for independent binomal distribution stratified by baseline severity; Proportion difference = 5.2, 90% CI 2-sided [-4.2 to 14.5]
Statistical Analysis 5: Comparison: Placebo vs Telcagepant 280 mg; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for independent binomal distribution stratified by baseline severity; Proportion difference = 34.7, 90% CI 2-sided [25.3 to 43.4]

3. Primary Outcome: Number of Participants Experiencing Adverse Events Within 48 Hours Post-dose (Count ≥4 in One or More Treatment Groups)
Description: An adverse event is any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment.
Time Frame: Up to 48 hours post-dose
Population: All participants as treated (one participant assigned to the Telcagepant 280 mg arm only took the placebo tablet and is included in the Placebo arm for adverse event reporting).
Measure: Number; unit: Participants
Arm/Group | Placebo | Telcagepant 280 mg +Ibuprofen 400 mg | Telcagepant 280 mg +APAP 1000 mg | Telcagepant 280 mg
Number analyzed (Participants) | 148 | 145 | 133 | 137
Participants | 27 | 44 | 42 | 34

4. Primary Outcome: Number of Participants Experiencing Adverse Events Within 14 Days Post-dose (Count ≥4 in One or More Treatment Groups)
Description: as for outcome 3
Time Frame: Up to 14 days post-dose
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | Telcagepant 280 mg +Ibuprofen 400 mg | Telcagepant 280 mg +APAP 1000 mg | Telcagepant 280 mg
Number analyzed (Participants) | 148 | 145 | 133 | 137
participants | 31 | 46 | 46 | 37

ADVERSE EVENTS:
Time Frame: Up to 14 days after the dose was taken.
Description: One participant randomly assigned to the Telcagepant 280 mg arm took only the placebp tablet and is included in the Placebo arm for adverse event reporting.
Arm/Group | Placebo | Telcagepant 280 mg +Ibuprofen 400 mg | Telcagepant 280 mg +APAP 1000 mg | Telcagepant 280 mg
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/145 | 0/133 | 0/137
Other Adverse Events (participants affected / at risk) | 12/148 | 23/145 | 16/133 | 16/137
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=148) | Telcagepant 280 mg +Ibuprofen 400 mg (N=145) | Telcagepant 280 mg +APAP 1000 mg (N=133) | Telcagepant 280 mg (N=137)
Nausea (Gastrointestinal disorders) | 8 (8) | 9 (9) | 5 (5) | 6 (6)
Fatigue (General disorders) | 1 (1) | 8 (9) | 7 (7) | 4 (4)
Somnolence (Nervous system disorders) | 3 (3) | 8 (8) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.